CLINICAL TRIAL: NCT06046781
Title: The Necessity and Timing of Exercise After Lumbar Disc Herniation Surgery: A Randomized Controlled Trial
Brief Title: Exercise After Lumbar Disc Herniation Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Safak Cine, MD, Istanbul Medeniyet University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SC/2023
Record Dates: First submitted 2023-09-13; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Disc Herniation; Surgery
Keywords: Lumbar disc herniation; Lumbar microdiscectomy; physical exercise
MeSH Terms: conditions — Intervertebral Disc Displacement; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: A total of 204 patients who underwent surgery for lumbar disc herniation were included and subsequently randomized into five groups. One group served as the control and was advised not to participate in any postoperative exercise. The remaining groups were recommended different exercises, which began at various times after surgery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Control group (Other): One group served as the control and was advised not to participate in any postoperative exercise.
  Interventions: Other: physical exercise
- Second week walking group (Experimental): Postoperative walking initiated 2 weeks following surgery.
  Interventions: Other: physical exercise
- One month walking group (Experimental): Postoperative walking initiated one month following surgery.
  Interventions: Other: physical exercise
- Second week waist exercise group (Experimental): Postoperative waist exercise initiated 2 weeks following surgery.
  Interventions: Other: physical exercise
- One month waist exercise group (Experimental): Postoperative waist exercise 1 month following surgery.
  Interventions: Other: physical exercise

INTERVENTIONS:
Other: physical exercise — The patients were randomized into 5 groups as control group, walking at 2 weeks, walking at 4 weeks, waist exercise at 2 weeks, waist exercise at 4 weeks.

SUMMARY:
Physical therapy and rehabilitation may improve low back pain and quality of life after lumbar disc herniation. But there is not any agreement of its optimal start time, and rehabilitative methods. This study evaluates the effects of early and late rehabilitation to the low back pain and quality of life following unilateral microdiscectomy.

DETAILED DESCRIPTION:
Lumbar disc herniation (LDH) is a frequently encountered ailment in neurosurgery clinics and is prevalent among the general populace, with a reported incidence of about 2%. As it is primarily observed in the workforce, it adversely affects their quality of life. One common reason for referring a patient for surgery is radiculopathy and low back pain co-occurrence. LDH is typically observed in the adult population in active occupation. Most patients with LDH can be treated conservatively, but surgery may be necessary for around 13% of cases.

The decision to operate depends on the individual patient, but persistent radicular pain and neurological dysfunction unresponsive to conservative treatment are common indications. Minimally invasive surgical techniques are becoming more prevalent. Currently, microsurgery is the most common approach for lumbar disc herniation. In addition, endoscopic and minimally invasive surgeries have become more prevalent.

Lumbar microdiscectomy is a surgical procedure involving discectomy with paravertebral muscle dissection. Subsequently, patients may experience postoperative back pain, potentially impacting their quality of life. Physical rehabilitation is frequently suggested following surgery. Some studies have indicated that physical therapy and rehabilitation may not significantly improve low back pain and quality of life after lumbar disc herniation. There is yet to be an agreement on the effectiveness of physical therapy, its optimal start time, and rehabilitative methods.

This study evaluates the effects of early and late rehabilitation following unilateral microdiscectomy for lumbar disc herniation. It also examines the differences in low back pain and patients' quality of life due to exercise.

ELIGIBILITY:
Inclusion Criteria:

* radicular pain that persisted despite 4-6 weeks of conservative treatment,
* detection of single-level disc herniation in MRI lumbar microsurgery.
* Individuals who underwent single-level unilateral lumbar microsurgery. Those with a surgical incision <3 cm.

Exclusion Criteria:

* Individuals with more than one level of muscle exposure at the time of surgery.
* those with a skin incision >3 cm

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-07 (Actual)

PRIMARY OUTCOMES:
Affect on back pain | 0 - 1 Months in the post-operative period
  Different effects of early and late rehabilitation to the low back pain following unilateral microdiscectomy. Pain status will be evaluated with the Visual Analogue Scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medeniyet University Medical Faculty Goztepe Suleyman Yalcin City Hospital, Istanbul, Kadıkoy, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
The raw data could be shared for further experimental and statistics analysis purposes.

REFERENCES:
- [Background] Kim YK, Kang D, Lee I, Kim SY. Differences in the Incidence of Symptomatic Cervical and Lumbar Disc Herniation According to Age, Sex and National Health Insurance Eligibility: A Pilot Study on the Disease's Association with Work. Int J Environ Res Public Health. 2018 Sep 25;15(10):2094. doi: 10.3390/ijerph15102094. PMID 30257414
- [Background] Hlubek RJ, Mundis GM Jr. Treatment for Recurrent Lumbar Disc Herniation. Curr Rev Musculoskelet Med. 2017 Dec;10(4):517-520. doi: 10.1007/s12178-017-9450-3. PMID 29103156
- [Background] Huang W, Han Z, Liu J, Yu L, Yu X. Risk Factors for Recurrent Lumbar Disc Herniation: A Systematic Review and Meta-Analysis. Medicine (Baltimore). 2016 Jan;95(2):e2378. doi: 10.1097/MD.0000000000002378. PMID 26765413
- [Background] Lewis RA, Williams NH, Sutton AJ, Burton K, Din NU, Matar HE, Hendry M, Phillips CJ, Nafees S, Fitzsimmons D, Rickard I, Wilkinson C. Comparative clinical effectiveness of management strategies for sciatica: systematic review and network meta-analyses. Spine J. 2015 Jun 1;15(6):1461-77. doi: 10.1016/j.spinee.2013.08.049. Epub 2013 Oct 4. PMID 24412033
- [Background] Rasouli MR, Rahimi-Movaghar V, Shokraneh F, Moradi-Lakeh M, Chou R. Minimally invasive discectomy versus microdiscectomy/open discectomy for symptomatic lumbar disc herniation. Cochrane Database Syst Rev. 2014 Sep 4;2014(9):CD010328. doi: 10.1002/14651858.CD010328.pub2. PMID 25184502
- [Background] Yoon SM, Ahn SS, Kim KH, Kim YD, Cho JH, Kim DH. Comparative Study of the Outcomes of Percutaneous Endoscopic Lumbar Discectomy and Microscopic Lumbar Discectomy Using the Tubular Retractor System Based on the VAS, ODI, and SF-36. Korean J Spine. 2012 Sep;9(3):215-22. doi: 10.14245/kjs.2012.9.3.215. Epub 2012 Sep 30. PMID 25983818
- [Background] Parker SL, Mendenhall SK, Godil SS, Sivasubramanian P, Cahill K, Ziewacz J, McGirt MJ. Incidence of Low Back Pain After Lumbar Discectomy for Herniated Disc and Its Effect on Patient-reported Outcomes. Clin Orthop Relat Res. 2015 Jun;473(6):1988-99. doi: 10.1007/s11999-015-4193-1. PMID 25694267
- [Background] Hebert JJ, Fritz JM, Thackeray A, Koppenhaver SL, Teyhen D. Early multimodal rehabilitation following lumbar disc surgery: a randomised clinical trial comparing the effects of two exercise programmes on clinical outcome and lumbar multifidus muscle function. Br J Sports Med. 2015 Jan;49(2):100-6. doi: 10.1136/bjsports-2013-092402. Epub 2013 Sep 12. PMID 24029724
- [Background] Barbosa TP, Raposo AR, Cunha PD, Cruz Oliveira N, Lobarinhas A, Varanda P, Direito-Santos B. Rehabilitation after cervical and lumbar spine surgery. EFORT Open Rev. 2023 Aug 1;8(8):626-638. doi: 10.1530/EOR-23-0015. PMID 37526242
- [Result] Vialle LR, Vialle EN, Suarez Henao JE, Giraldo G. LUMBAR DISC HERNIATION. Rev Bras Ortop. 2015 Nov 16;45(1):17-22. doi: 10.1016/S2255-4971(15)30211-1. eCollection 2010 Jan. PMID 27019834